













MEXICAN SOCIAL SECURITY INSTITUTE
EDUCATION, RESEARCH AND HEALTH POLICY UNIT
HEALTH RESEARCH COORDINATION
HIGH SPECIALTY MEDICAL UNIT (UMAE) "DR. BERNARDO SEPÚLVEDA"
CENTRO MÉDICO NACIONAL SIGLO XXI, IMSS, CDMX.
MEDICAL RESEARCH UNIT IN BIOCHEMISTRY.
DEPARTMENT OF NEUROLOGY AND NEUROPHYSIOLOGY.
FAMILY MEDICINE UNITS NUMBER 20, 41 AND 44, IMSS, CDMX.
SPECIALTY OF HUMAN ACUPUNCTURE OF THE ENMH OF THE IPN

## Official Title of the study:

"Evaluation of the effect of electroacupuncture on the sensory symptoms of Symmetrical Distal Polyneuropathy of Diabetic origin and its correlation with changes in Nerve Conduction Velocity."

MEXICAN SOCIAL SECURITY INSTITUTE AND EDUCATION, RESEARCH AND HEALTH POLICY UNIT STUDY VERIFICATION ID: R-2020-785-070.

CONBIOÉTICA-09-CEI-009-20160601.

NCT Number: NOT AVAILABLE.

DOCUMENT OF APPROVAL OF THE RESEARCH PROTOCOL.

DATE: May 26th, 2020.



## Dirección de Prestaciones Médicas Unidad de Educación, Investigación y Politicas de Salud Coordinación de Investigación en Salud



## Dictamen de Aprobación

Martes, 26 de mayo de 2020

Ref. 09-B5-61-2800/202000/

Dr. JOSE DE JESUS PERALTA ROMERO Unidad de Investigación Médica en Bioquímica Siglo XXI (U INVEST MED EN BIOQUIM S XXI) Nivel Central

Presente:

Informo a usted que el protocolo titulado: EVALUACIÓN DEL EFECTO DE LA ELECTROACUPUNTURA EN LOS SÍNTOMAS SENSITIVOS DE LA POLINEUROPATÍA DISTAL SIMÉTRICA DE ORIGEN DIABÉTICO Y SU CORRELACIÓN CON CAMBIOS EN LA VELOCIDAD DE CONDUCCIÓN NERVIOSA, fue sometido a la consideración de este Comité Nacional de Investigación Científica.

Los procedimientos propuestos en el protocolo cumplen con los requerimientos de las normas vigentes, con base en las opiniones de los vocales del Comité de Ética en Investigación y del Comité de Investigación del Comité Nacional de Investigación Científica del IMSS, se ha emitido el dictamen de **APROBADO**, con número de registro: R-2020-785-070.

De acuerdo a la normatividad vigente, deberá informar a esta Comité en los meses de enero y julio de cada año, acerca del desarrollo del proyecto a su cargo. Este dictamen sólo tiene vigencia de un año. Por lo que en caso de ser necesario requerirá solicitar una reaprobación al Comité de Ética en Investigación del Comité Nacional de Investigación Científica, al término de la vigencia del mismo.

Atentamente,

Dra. María Susana Navarrete Navarro

Secretaria Ejecutiva

Comité Nacional de Investigación Científica

Anexo comentarios: Se anexa dictamen

SNN/ iah. F-CNIC-2019-068

**IMSS**